CLINICAL TRIAL: NCT02885688
Title: Early Metabolic Support as a Potential Solution to Multi-Organ Dysfunction Syndrome (MODS) During Severe Sepsis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-1014
Record Dates: First submitted 2016-08-17; First posted 2016-08-31 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Septic Shock
Keywords: Septic Shock; Sepsis; Standard of care; Liquid nutrition; Metabolic support; Enteral nutrition; Insulin Drip; Glucose Drip
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard-of-Care Treatment for Sepsis (Other): Participants with diagnosis of septic shock in MD Anderson Cancer Center ICU receive standard of care treatment alone for up to 7 days.
  Interventions: Procedure: Insulin Drip
- Standard-of-Care Treatment Plus Liquid Nutrition for Sepsis (Experimental): Participants with diagnosis of septic shock in MD Anderson Cancer Center ICU receive standard of care treatment plus plus liquid nutrition for up to 7 days.
  Interventions: Dietary Supplement: Liquid Nutrition; Procedure: Insulin Drip

INTERVENTIONS:
Dietary Supplement: Liquid Nutrition — Participants receive liquid nutrition by vein non-stop for up to 7 days.
  Other Names: Metabolic support; Enteral nutrition
  Arms: Standard-of-Care Treatment Plus Liquid Nutrition for Sepsis
Procedure: Insulin Drip — Insulin drip by vein to keep serum glucose level between 140 and 180 mg/dL as per ICU protocol.
  The interventions required in the current standard management of patients with septic shock is based on the MD Anderson Evidence-Based Protocol (EBP) for management of Severe Sepsis initiated on admission to the ICU.
  Other Names: Glucose Drip

SUMMARY:
The goal of this clinical research study is to learn if adding liquid nutrition therapy that is given by vein to standard-of-care treatment for sepsis can help to control sepsis symptoms better than giving standard-of-care treatment alone.

Researchers also want to compare the length of ICU and hospital stay and any side effects between these 2 treatments.

DETAILED DESCRIPTION:
Study Groups and Procedures:

If participant is eligible and chooses to take part in this study, they will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

Group 1 will receive standard-of-care treatment alone for up to 7 days.

Group 2 will receive standard treatment for up to 7 days, plus liquid nutrition. The liquid nutrition will be given by vein non-stop for up to 7 days. The liquid nutrition therapy may stop sooner if participant's doctor thinks they are ready, based on how they are tolerating tube feeding.

Both Groups: As part of standard treatment, participants will receive breathing and blood pressure support, daily routine blood draws, imaging, standard drugs (such as antibiotics and blood pressure drugs), and other tests the doctor decides are needed. These tests and treatment will begin within 12 hours after participant is admitted to the ICU.

Participant's doctor will discuss the standard treatment and tests with them in more detail. Participant may ask the study staff for information about how the standard treatment and tests are given and their risks.

If participant is in Group 2, blood (about 4 teaspoons) will be drawn on Days 1-7 to check their blood oxygen and sugar levels. These tests may help the doctor make any needed changes to participant's liquid nutrition therapy.

Length of Participation:

Participant will take part in this study for up to 7 days. Patient's participation on this study will be over after Day 7 or when they can leave the ICU, whichever happens first. Participant may be taken off study early if intolerable side effects occur or if they are unable to follow study directions.

This is an investigational study. The liquid nutrition provided in this study is FDA approved and commercially available. Comparing the 2 study groups is investigational. The study doctor can explain how the liquid nutrition is designed to work.

Up to 50 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All adult patients 18-years-old or greater
2. Admitted to the adult medical intensive unit (MICU) of MD Anderson Cancer Center
3. Diagnosis of Sepsis within 12 hours of MICU admission defined as: 1) Suspected or documented infection and 2) Acute increase of >/= 2 SOFA points (a proxy for organ dysfunction)
4. Diagnosis of Septic Shock within 12 hours of MICU admission defined as meeting criteria for sepsis (see inclusion criteria C) in addition to the following: 1) Vasopressor therapy needed to elevate MAP >/= 65 mmg Hg and 2) Lactate > 2 mmol/L (18 mg/dL) after adequate fluid resuscitation
5. Sequential Organ Failure Assessment (SOFA) score meeting the following requirements: 1) Cardiovascular SOFA >/= 2 and 2) Total SOFA score of less than 15
6. Diagnosis of leukemia, lymphoma, or status post stem cell transplantation
7. Patients in septic shock and not able to tolerate enteral nutrition above 70 percent of their daily nutritional caloric intake.

Exclusion Criteria:

1. Children (patients < 18-years-old) of age are not admitted to the MICU but to the pediatric intensive care unit (PICU)
2. Do Not Resuscitate (DNR), Comfort Care or Moribund
3. Death expected within the next 24 hours
4. Active Bleeding
5. End-stage Renal Disease (ESRD)
6. Chronic Liver Disease: Childs-Pugh Class C and/or Diagnosis of Cirrhosis
7. Tumor Lysis Syndrome
8. Sulfite Allergy: Hepatamine contraindicated. More common in asthmatics. (Please note that this is NOT sulfa allergy and is NOT contraindicated in patients with sulfa allergy)
9. Serum sodium concentration < 130 milliequivalent (mEq)/L or >150 mEq/L (Note: Once serum sodium levels are >/= 130 or </= 150 mEq/L within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.)
10. Serum Creatinine level: SCr > 2.5 mg/dL (Note: Once serum creatinine levels are =/< 2.5 mg/dL within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.)
11. 11) Urine output < 400 cc/24hrs (Note: Once urine output levels are >/= 400 cc within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.)
12. Hyperkalemia K > 5.5 mEq/L (Note: Once potassium levels are </= 5.5 mEq/L within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.)
13. Hyperglycemia: Glucose > 250 mg/dL (Note: Once glucose is </= 250 mg/dL within 12 hours after meeting inclusion criteria, the patient can then be considered for the study. This is only a temporary restriction.)
14. Hyperphosphatemia: Serum Phosphorous > 8.0 mg/dL
15. Patient with a history of metabolic abnormality in any one of the following amino acids: Alanine, Arginine, Cysteine hydrochloride, Glycine, Histidine, Isoleucine, Leucine, Lysine acetate, Methionine, Phenylalanine, Phosphoric ac-id, Proline, Serine, Threonine, Tryptophan, and Valine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Early Metabolic Support in Participants with Sepsis Determined by Accrual | 7 days
  Trial feasible if ≥ 50% of eligible patients consent (i.e., approach 100 patients to achieve 50 that consent).
Feasibility of Early Metabolic Support in Participants with Sepsis Determined by Adherence | 7 days
  Trial feasible if ≥ 60% of enrolled patients complete the treatments up to 7 days or upon discharge from the ICU, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Diego de Villalobos, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org